CLINICAL TRIAL: NCT05326360
Title: The Effect of Additional Administration of Ramosetron on Late PONV (Postoperative Nausea and Vomiting) in Patients Undergoing Breast Surgery
Brief Title: Ramosetron on Late PONV (Postoperative Nausea and Vomiting)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Eunsoo Kim, Associate professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012-001-108
Record Dates: First submitted 2022-03-16; First posted 2022-04-13 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Nausea and Vomiting; Breast Cancer Female
Keywords: mastectomy; postoperative nausea and vomiting; ramosetron
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group C (No Intervention): receive ramosetron i.v. 0.3mg at the end of surgery without additional ramosetron
- group B (Experimental): receive ramosetron i.v. 0.3mg at the end of surgery with two additional doses of ramosetron at 12- and 24- hour postoperative time points
  Interventions: Drug: Ramosetron Hydrochloride
- group M (Experimental): receive ramosetron i.v. 0.3mg at the end of surgery followed ramosetron 0.6 mg mix with the patient-controlled analgesia (PCA) regimen
  Interventions: Drug: Ramosetron Hydrochloride

INTERVENTIONS:
Drug: Ramosetron Hydrochloride — we injected two additional remosetron doses in different way in experimental groups. In group B, patients received additional ramosetron at 12 hour interval, in group M, patients received additional ramosetron in mixed with the patient controlled analgesia regimen.
  Arms: group B; group M

SUMMARY:
The purpose of this study was to evaluate the effectiveness of additional ramosetron injection for controlling late postoperative nausea and vomiting (PONV) after breast surgery in high risk PONV patients. The investigators compared PONV amomng 3 groups- group C: no additional ramosteron, group B: two additional ramosteron doses at 12 hour interval, group M: two additional ramosetron doses mix to the intraveonus patient controlled analgesia.

DETAILED DESCRIPTION:
The investigators included high risk patients of PONV with a score of 3 or more as measured by the Apfel's score and over 18 years old who receive breast surgery and intravenous patient controlled analgesia. All patients was received ramosetron 0.3 mg at the end of surgery. The patients were evaluated for number of PONV (nausea, vomiting, retching) at 1, 6, 24, and 48 hours postoperatively. Nausea was defined as an unpleasant feeling of vomiting. Retching was defined as an excessive contraction or a regular movement. of the respiratory muscles where no gastric contents were excreted, and vomiting was defined as the excretion of gastric contents. PONV were further detailed quantified using the RINVR score (Rhodes Index of Nausea, Vomiting, and Retching) which enabled the patients' objective and subjective symptoms to be evaluated as a simple and reliable methods.

Intravenous injection of ondansetron 4 mg was administered as a rescue antiemetic. The patients were evaluated 2 hours after ondansetron administration. If the symptom persisted, use of second rescue antiemetics dexamethasone 5 mg.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* American Society of Anesthesiologists (ASA) physical status I or II
* requesting IV PCA (patient control of analgesia) for pain control
* the high-risk group of PONV with a score of 3 or more as measured by the Apfel's score.

Exclusion Criteria:

* emergency operation
* re-operation
* drug abuse, allergy
* major organ disease (gastrointestinal, cardiovascular, respiratory, cerebral, renal or hepatic disease)
* smoker
* pregnancy
* lactation
* previously use of antiemetics or systemic steroids within 48 before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
number of PONV | 24hour postoperatively
  number of nausea, vomiting, retching

SECONDARY OUTCOMES:
number of PONV | 1hour, 6hour, 48 hour postoperatively
  number of nausea, vomiting, retching
Rhodes Index of Nausea, Vomiting, and Retching (RINVR) score | 1hour, 6hour, 24hour, 48 hour postoperatively
  further detaied quantified in PONV experience, total score: 32, none:0, mild: 1-8 point, moderate: 9-16 point, great: 17-24 point, severe: 25-32 point

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hopsital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided